CLINICAL TRIAL: NCT06174467
Title: Learning for Hearts and Minds (ACM) in Elementary School Students From Public Schools: a Randomized Controlled Trial on Socio-emotional Skills and Brain Functioning
Brief Title: Learning for Hearts and Minds in Elementary School
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Emory University (Other); Gaia Mais (Unknown); Universidade Federal do ABC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ACM-Students-Intervention
Record Dates: First submitted 2023-02-24; First posted 2023-12-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-02

CONDITIONS: Social Emotional Learning
Keywords: learning; social-emotional learning; emotion regulation; prosocial behavior
MeSH Terms: conditions — Emotional Regulation; Altruism

STUDY DESIGN:
Intervention Model Description: Elementary school students from public schools (N = 600) will be invited to participate in the Learning for Hearts and Minds Training.
  Inclusion criteria: being students of the 4th and 5th years of elementary school I.
  Exclusion criteria: not having both terms signed (free and informed consent by those responsible and assent by the students). The student is undergoing neurological or psychiatric treatment (in this case, students will be invited to participate in the training, but will not be included in the study sample). The teacher responsible for the classroom is undergoing neurological or psychiatric treatment, or has a condition that prevents him from applying the TACM. The teacher in charge did not sign the free and informed consent form for their participation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First group to receive the intervention (Experimental): This cluster of classes of different scholls will be instructed in the social emotional and ethical learning training (SEELearning) and being tested trought questionaries.
  Interventions: Behavioral: SEELearning Training
- Second group to receive the intervention (Experimental): The cluster of classes of different scholls forming the second group, will not be instructed in the social emotional and ethical learning training (SEELearning) in the first semester, but will answer the questionaries during this period. Than, in next semester they will receive the Training.
  Interventions: Behavioral: Waiting list group of the intervention

INTERVENTIONS:
Behavioral: SEELearning Training — This group will receive the Learning Training for Hearts and Minds and will be submitted to assessments and questionnaires that measure the improvement of well-being, reduction of stress and literacy in the contents and human values taught in the training.
  The program aims to increase participants' awareness, compassion and engagement. Compassion refers to cultivating a way of relating to oneself, others and humanity through kindness, empathy and genuine care for the happiness and suffering of these individuals. Awareness refers to cultivating a detailed, first-person understanding of thoughts, feelings, and emotions.
  Arms: First group to receive the intervention
Behavioral: Waiting list group of the intervention — The group will remain on a waiting list and will respond to questionnaires about well-being and other items before receiving the training and, in the second semester, during the period in which it will receive the training
  Arms: Second group to receive the intervention

SUMMARY:
ABSTRACT- Introduction: Skills such as recognizing and managing emotions, developing empathy, building cooperative relationships, solving problems effectively and obtaining communication skills have gained importance in several schools and this has been made possible by Socio-Emotional Learning (SEL). Robust studies in this area in Latin America are lacking, and what happens in the brain and in our general physiology, from trainings related to SEL, needs to be better understood. Objectives: To assess the effects of Learning for Hearts and Minds Training (TACM) on positive and negative affect, empathy and compassion, emotional expression, self-compassion, life satisfaction, sense of community in the classroom, academic goals, school performance, brain activity and heart rate variability in 4th and 5th year elementary school students. Methods: This is a randomized controlled trial in clusters with cross-over, in approximately 600 students. By the end of the first semester, one group of students will receive the TACM and the other will be a waiting control group. In the second semester, the latter will receive the TACM and the former will continue the TACM practices. The groups will be evaluated in 5 moments during the year. A classroom will be randomly assigned to undergo an assessment of brain activity and cardiac variability to assess their ability to regulate emotions. Students, parents and teachers will be drawn for a qualitative interview at the end of the academic semesters about the effects of TACM.

ELIGIBILITY:
Inclusion Criteria:

* Students of selected public schools of Junidaí of the 4th and 5th grade of Brazilian elementary School

Exclusion Criteria:

-

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-12-17 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and negative Affects scores | 1 year
  they will answer the "Positive and Negative Affect Scale for Children (PANAS-C) questionary." Consisting of 34 items, with 17 items in each subscale, it is used to measure children's emotions during the previous weeks. The subscales measure positive and negative affect. The scale features words that describe different feelings and emotions on a 5-item Likert scale, ranging from 1 ("very little or not at all") to 5 ("extremely").
Change in Empathy and Compassion | 1 year
  Students will respond to the "Empathy and Compassion Scale" Consisting of 14 items, it assesses empathy and the ability to take perspective. It assesses how the individual relates to the difficulties faced by other people. It features a 5-item Likert scale ranging from "not at all like me" to "exactly how I
Change in emotional expression scores | 1 year
  They will answer the "Emotional Expression Scale in Children" It presents 6 questions about the child's ability to express their emotions. Each question is answered on a 5-item Likert scale ranging from "not at all true" to "completely true".
Change in Self-compassion sco4es | 1 year
  They will answer the Self-Compassion Scale - short version It has 12 questions about how the individual treats himself compared to the way he treats other people. Each question is answered on a 5-item Likert scale ranging from "never" to "always".
Change in satisfaction with life perception scores | 1 year
  They will answer the Life Satisfaction Scale for Children It has 5 questions about how satisfied the child is with his life. The Likert scale has 5 items ranging from "totally disagree" to "totally agree"
Change in sense of comunity in the classroom scores | 1 year
  They will answer the Scale of Sense of Community in the Classroom The scale has 14 items that assess students' perception in the classroom as belonging to a community and promoting group values. The 5-item Likert scale ranges from "strongly disagree" to "strongly agree" .
Change in Academic Objectives scores | 1 year
  They will answer the Academic Objectives Scale Scale of 6 items in which the student states about his perception of achieving learning objectives. 5-point Likert scale ranges from "not at all like me" to "exactly like me".
the effects of TACM on students' ability to regulate their emotions by assessing their brain activity and cardiac variability | 1 year
  Groups of children who were submitted to TACM will be avaluated in their emotional regulation capacities and have their brain activities and cardiac variability measured by Fnears and Polar before in 2 moments (before the training just before the end of the first semester and near the end of the school year, when they have already received all the training TACM)
the effects of TACM on students' ability to regulate their emotions by assessing their brain activity | 1 year
  Groups of children who were submitted to TACM will be avaluated in their emotional regulation capacities and have their brain activities measured by FNIRS (functional near infrared spectroscopy) in 2 moments (before the training just before the end of the first semester and near the end of the school year, when they have already received all the training TACM)
Change in School performance | 1 year
  Classification of colleagues according to social characteristics:
  In this report, students will make lists of colleagues who have the following characteristics: students who are generous; who show compassion; who get along well with others; get along well with their teachers.
the effects of TACM on students' ability to regulate their emotions by assessing their heart rate variability the effects of TACM on student's ability to regulate their emotions by assessing the heart rate variability | 1 year
  We will measure the heart rate variability using a Polar belt

SECONDARY OUTCOMES:
Teachers TACM Literacy and aplication | 1 year
  The teachers responsible for the classrooms will be trained in TACM during the semester and will be evaluated in terms of attendance at training, filling out questionnaires, participating in chats, self-assessing their levels of stress, frustration, well-being, motivation and attention in a scale (items ranging from 0 to 10).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil